CLINICAL TRIAL: NCT03798236
Title: Randomized, Double Blind, Placebo Controlled "First-in-human" Study to Assess the Safety and Tolerability of Single Ascending Oral Doses of PBF-1650 (40 mg, 80 mg, 120 and 240 mg) in Healthy Young Male Volunteers.
Brief Title: Study to Assess the Safety and Tolerability of PBF-1650 in Healthy Volunteers.
Acronym: ADENOIMMUNE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Clínica Universidad de Navarra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PBF-1650CT-01
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Psoriasis
Keywords: Adenosine A3 receptor antagonist; autoimmune diseases; Immune modulator
MeSH Terms: conditions — Psoriasis; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, placebo-controlled clinical study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PBF-1650 40mg (Experimental)
  Interventions: Drug: PBF-1650 oral capsules
- PBF-1650 80mg (Experimental)
  Interventions: Drug: PBF-1650 oral capsules
- PBF-1650 120mg (Experimental)
  Interventions: Drug: PBF-1650 oral capsules
- PBF-1650 240mg (Experimental)
  Interventions: Drug: PBF-1650 oral capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: PBF-1650 oral capsules — Adenosine A3 receptor (AA3R) antagonist
  Arms: PBF-1650 120mg; PBF-1650 240mg; PBF-1650 40mg; PBF-1650 80mg
Drug: Placebo oral capsule — solid microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Single center, randomized, double-blind, placebo-controlled clinical study to assess the safety and tolerability of PBF-1650 in order to obtain the Maximum Tolerated Dose (MTD).

DETAILED DESCRIPTION:
The clinical trial will be a dose escalation study without therapeutic benefit, in which PBF-1650 will be administered as single oral ascending- dose to healthy young male volunteers. Up to four different rising doses will be tested (40 mg, 80 mg, 120 and 240 mg) in groups/cohorts of 8 participants. Thus, four groups/cohorts will participate. For each dose level / group, the participants will be randomized to active or placebo with 2 participants being randomly assigned to placebo and 6 to the active drug. First, one volunteer will receive active drug (subgroup 1); after at least 48h of safety and tolerability assessment a second subgroup of 3 volunteers will receive 2 active drug and 1 placebo; after at least another 48h of safety and tolerability parameters assessment a third subgroup of 4 volunteers will receive 3 active drug and 1 placebo. After evaluation of safety parameters of corresponding dose level, the process will replicate one week afterwards in the following dosages.

The pharmacokinetics profile of PBF-1650 after single oral dose administration of the four dose levels will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18-45 years (inclusive) of age at the time of enrollment.
* Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner use some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
* Clinically acceptable blood pressure and pulse rate in supine and standing position (SBP between 140-100 mm Hg/ DBP between 90-50 mm Hg / HR between 100-50 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
* Body weight within normal range (Quetelet's index between 19 and 26) expressed as weight (kg) / height (m2).
* Able to understand the nature of the study and comply with all their requirements.
* Free acceptance to participate in the study by obtains signed informed consent form approved by the Ethics Committee (CEIm).

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* Background or clinical evidence of chronic diseases.
* Acute illness two weeks before drug administration.
* Having undergone major surgery during the previous 6 months.
* Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication).
* History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 g or high consumption of stimulating beverages (> 5 coffees, teas or coca cola drinks/ day).
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Need of any prescription medication within 14 days prior to the administration of the investigational drug and non-prescription medication or herbal medicines within 7 days prior to the administration of the drug. Paracetamol (acetaminophen) is allowed, at doses up to 1 g daily, at the investigator discretion.
* Participation in other clinical trials during the previous 90 days in which an investigational drug or a commercially available drug was tested.
* Having donated blood during 3 months' period before inclusion in the study.
* Existence of any surgical or medical condition which might interfere with the absortion, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract
* 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradychardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
* Symptoms of a significant somatic or mental illness in the four-week period preceding drug administration.
* History of hepatitis HBV and / or HCV and / or positive serology results, which indicate the presence of hepatitis B surface antigen and / or detectable HCV ribonucleic acid (RNA).
* Positive results from the HIV serology.
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation.
* Positive results of the drugs at screening period or the day before starting treatment period. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the Principal Investigator).
* Known hypersensitivity to the study drug or the composition of the galenical form.
* History of psychiatric diseases or epileptic seizures.
* Pill swallowing difficulties.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | 7 Days
  Adverse Events will be qualified according to the definitions and values stated in CTCAE V04 v4)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain